CLINICAL TRIAL: NCT05411783
Title: Low Tie Versus High Tie of the Inferior Mesenteric Vein During Colorectal Cancer Surgery: A Randomized Clinical Trial. LOTHVEIN Study
Brief Title: Low Tie Versus High Tie of the Inferior Mesenteric Vein During Colorectal Cancer Surgery: A Randomized Clinical Trial
Acronym: LOTHVEIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Carlo di Nancy Hospital (Other)
Responsible Party: Principal Investigator, Giovanni Guglielmo Laracca, MD, San Carlo di Nancy Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LOTHVEIN
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Anastomotic Leak; Anastomotic Leak Large Intestine; Anastomotic Leak Rectum; Colon Cancer; Colon Neoplasm; Rectum Cancer; Rectum Neoplasm; Colorectal Cancer
Keywords: colorectal surgery; IMV tie; anastomotic leak
MeSH Terms: conditions — Anastomotic Leak; Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High tie of IMV (No Intervention): The IMV will be tie under the pancreas as the usual procedure in left hemicolectomy and ARR
- Low tie of IMV (Experimental): The IMV will be tie under the left colic vein
  Interventions: Procedure: Low tie of IMV

INTERVENTIONS:
Procedure: Low tie of IMV — The IMV will be tie under the left colic vein
  Arms: Low tie of IMV

SUMMARY:
This study aim to determine if a different surgical technique could result in a lower anastomotic leak rate. The two techniques are equally used around the world and well described by the international literature but this is the first study that compare the two techniques.

DETAILED DESCRIPTION:
Colorectal cancer accounts for approximately 10% of all annually diagnosed cancers and cancer-related deaths worldwide. It is the second most common cancer diagnosed in women and third most in men. In women, incidence and mortality are approximately 25% lower than in men. These rates also vary geographically, with the highest rates seen in the most developed countries. With continuing progress in developing countries, the incidence of colorectal cancer worldwide is predicted to increase to 2·5 million new cases in 2035. Stabilising and decreasing trends tend to be seen in highly developed countries only. These have been primarily attributed to nationwide screening programmes and increased uptake of colonoscopy in general, although lifestyle and dietary changes might also contribute. In contrast, a worrying rise in patients presenting with colorectal cancer younger than 50 years has been observed, especially rectal cancer and left-sided colon cancer. Although genetic, lifestyle, obesity, and environmental factors might have some association, the exact reasons for this increase are not completely understood.

The safety of colorectal surgery for oncological disease has dramatically improved over the last 50 years due to a better preoperative preparation, antibiotic prophylaxis, surgical technique, and postoperative management. Since abdomino-perineal resection, new and less aggressive procedures have been developed (e.g., laparoscopic and robotic approach, endoluminal resection), always respecting the concepts of oncologically free margins (R0) and of avoiding the dissemination of cancer cells during surgery. Several years ago, a further step forward in the field of colorectal surgery was the introduction of surgical stapler, which allowed surgeons to perform safer and quicker anastomoses especially during minimally invasive surgery. Moreover, in the last decades there has been a spread of minimal invasive procedures such as the total trans-anal mesorectal excision with an even better clinical outcome for the patients. There has also been the development and spread of robotic devices to aid surgical procedures.

However, complications after colorectal surgery are still inevitable. Their severity is variable ranging from mild with a minimal impact on the patient, to severe and potentially fatal, in case of anastomotic leak (AL). AL is one of the most severe complications for colorectal surgery owing to its negative impact on both short- and long-term outcomes. The incidence reported in the literature has not significantly changed in recent decades despite constant improvements in both stapled and manual sutures, in the pre-operative assessment of the patient, as well as in the surgical technique. The reported incidence is about 2.8-30% as all, of which 75% occurs in rectal anastomosis resulting in a mortality rate of 2-16.4% and in a morbidity rate of 20-35%. Many risk factors have been identified in association with AL, such as low-level anastomosis, male gender, and smoking; however, these factors are all patient-related and not modifiable. Among the other important elements more directly related to the surgeon's experience that can impair anastomotic healing, the most important are undue tension at the level of the anastomosis; technical failure of the stapler; insufficient blood perfusion. It is generally accepted that adequate perfusion is required for anastomotic healing and surgeons usually perform different checks before and after the completion of anastomosis. In fact, poor arterial vascularity is an independent predictor of anastomotic failure after rectal resection with colorectal anastomosis. Currently, there are no data about the role of the venous ischemia in AL. The tie of the inferior mesenteric vein (IMV) under the pancreas, is considered the standard, and it permits to reduce the tension on the anastomosis lengthening the colon segment. Some authors arguing that the high tie of the IMV is responsible for the venous stasis and the venous ischemia responsible for the AL. At present time doesn't exist any study that compare different level of IMV tie and the correlation with AL.

ELIGIBILITY:
Inclusion Criteria:

* Adenoma or adenocarcinoma of left colon or upper rectum without neoajuvant RCT
* No distant metastasis

Exclusion Criteria:

* Previous colonic surgery
* emergency surgery
* Previous pelvic radiation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leak | 30 day
  Anastomotic leak clinically or radiologically evident

SECONDARY OUTCOMES:
Post-operative complications | 30 day
  Any post-operative complication

CONTACTS AND LOCATIONS:
Locations (1):
- San Carlo di Nancy Hospital, Roma, RM, Italy

REFERENCES:
- [Background] Johdi NA, Sukor NF. Colorectal Cancer Immunotherapy: Options and Strategies. Front Immunol. 2020 Sep 18;11:1624. doi: 10.3389/fimmu.2020.01624. eCollection 2020. PMID 33042104
- [Background] Chiarello MM, Fransvea P, Cariati M, Adams NJ, Bianchi V, Brisinda G. Anastomotic leakage in colorectal cancer surgery. Surg Oncol. 2022 Mar;40:101708. doi: 10.1016/j.suronc.2022.101708. Epub 2022 Jan 24. PMID 35092916
- [Background] De Nardi P, Elmore U, Maggi G, Maggiore R, Boni L, Cassinotti E, Fumagalli U, Gardani M, De Pascale S, Parise P, Vignali A, Rosati R. Intraoperative angiography with indocyanine green to assess anastomosis perfusion in patients undergoing laparoscopic colorectal resection: results of a multicenter randomized controlled trial. Surg Endosc. 2020 Jan;34(1):53-60. doi: 10.1007/s00464-019-06730-0. Epub 2019 Mar 21. PMID 30903276
- [Background] Rojas-Machado SA, Romero-Simo M, Arroyo A, Rojas-Machado A, Lopez J, Calpena R. Prediction of anastomotic leak in colorectal cancer surgery based on a new prognostic index PROCOLE (prognostic colorectal leakage) developed from the meta-analysis of observational studies of risk factors. Int J Colorectal Dis. 2016 Feb;31(2):197-210. doi: 10.1007/s00384-015-2422-4. Epub 2015 Oct 27. PMID 26507962
- [Background] Boyle NH, Manifold D, Jordan MH, Mason RC. Intraoperative assessment of colonic perfusion using scanning laser Doppler flowmetry during colonic resection. J Am Coll Surg. 2000 Nov;191(5):504-10. doi: 10.1016/s1072-7515(00)00709-2. PMID 11085730
- [Background] Girard E, Trilling B, Rabattu PY, Sage PY, Taton N, Robert Y, Chaffanjon P, Faucheron JL. Level of inferior mesenteric artery ligation in low rectal cancer surgery: high tie preferred over low tie. Tech Coloproctol. 2019 Mar;23(3):267-271. doi: 10.1007/s10151-019-01931-0. Epub 2019 Apr 8. PMID 30963345
- [Background] Bonnet S, Berger A, Hentati N, Abid B, Chevallier JM, Wind P, Delmas V, Douard R. High tie versus low tie vascular ligation of the inferior mesenteric artery in colorectal cancer surgery: impact on the gain in colon length and implications on the feasibility of anastomoses. Dis Colon Rectum. 2012 May;55(5):515-21. doi: 10.1097/DCR.0b013e318246f1a2. PMID 22513429
- [Background] Graf O, Boland GW, Kaufman JA, Warshaw AL, Fernandez del Castillo C, Mueller PR. Anatomic variants of mesenteric veins: depiction with helical CT venography. AJR Am J Roentgenol. 1997 May;168(5):1209-13. doi: 10.2214/ajr.168.5.9129413.
- [Background] Garcia-Granero A, Pellino G, Frasson M, Primo Romaguera V, Fletcher-Sanfeliu D, Blasco Serra A, Valverde-Navarro AA, Martinez-Soriano F, Garcia-Granero E. Possible effects of height of ligation of the inferior mesenteric vein on venous return of the colorectal anastomosis: the venous trunk theory. Tech Coloproctol. 2019 Aug;23(8):799-800. doi: 10.1007/s10151-019-02038-2. Epub 2019 Jul 18. No abstract available. PMID 31321633